CLINICAL TRIAL: NCT07093944
Title: Effect of N-acetyl Cysteine as an Adjuvant Therapy on Symptoms and Progression of Parkinson's Disease
Brief Title: Randomized, Placebo-Controlled Trial of N-acetylcysteine In Parkinson's Disease Patients: A Pilot Study
Acronym: IRANNACPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kurdistan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arman Rahimmi, Assistant Professor, Kurdistan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.MUK.REC.1397/348; MUKIRAN (Other: Kurdistan University of Medical Sciences)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease; N-acetylcysteine
MeSH Terms: interventions — Acetylcysteine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded clinical trial study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication group (Experimental): Receiving 1200 mg N-acetylcysteine per day, twice daily, each time 600 mg
  Interventions: Drug: N-Acetylcysteine (NAC) Treatment
- Placebo group (Placebo Comparator): Receiving a placebo with similar appearance, color, odor, and taste like real medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) Treatment — Parkinson's disease patients receive NAC (1200 mg/day) for one year.
  Other Names: NAC; Fluimucil effervescent tablet
  Arms: Medication group
Drug: Placebo — Parkinson's disease patients receive Placebo similar to the real drug, with no active ingredient
  Arms: Placebo group

SUMMARY:
This is a study on Parkinson's disease patients, referred to Tohid Hospital of Sanandaj City. The patients receive N-acetylcysteine for one year. The efficacy of the Drug is evaluated based on clinical interview, filling Unified Parkinson's Disease Rating Scale (UPDRS) questionnaire, and single-photon emission computerized tomography (SPECT) brain imaging. The only person who has not been blinded for the study is the supplier of the drug and placebo.

Inclusion criteria: Patient's informed consent Exclusion criteria: Having brain surgery within a year before the initiation of the intervention.

Medication group: receiving 1200 mg N-acetylcysteine per day, twice daily, each time 600 mg.

placebo group: receiving a placebo with similar appearance, color, odor, and taste like real medication.

DETAILED DESCRIPTION:
This is a randomized double-blinded clinical trial. Randomization method is based on making blocks with size of 4 people, to divide participants into two groups: intervention group (A) and control group (B). So that, we divide all participants to four-sample blocks, and we allocate the block's samples equally between the two groups (e.g. ABAB). This pattern is the same in all blocks. Participants, clinical caregivers, outcome evaluators and data analyzers are not aware whether the therapeutic regimens include the drug or placebo. only the main researcher and pharmacist are aware of nature of therapeutic regimen based on codes given to the drug and placebo packages, earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patient's informed consent No brain surgery in the patient's post medical history

Exclusion Criteria:

* having brain surgery within a year before starting the treatment period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
single-photon emission computerized tomography (SPECT) brain imaging | one year
  Also known as TRODAT scan or DaTscan, is a nuclear medicine imaging procedure that helps diagnose and evaluate Parkinson's disease by assessing the function of dopamine transporters in the brain. It specifically visualizes the dopaminergic system, which is affected in Parkinson's disease.
Unified Parkinson's Disease Rating Scale (UPDRS) | one year for each PD patient (at baseline and after one year)
  It is a questionnaire to assess the severity and progression of Parkinson's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Kurdistan University of Medical Sciences, Sanandaj, Kurdistan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided